CLINICAL TRIAL: NCT03958227
Title: Istanbul University, Faculty of Health Science, Division of Physiotherapy and Rehabilitation
Brief Title: Investigation The Efficacy of Manual Therapy and Exercise in Patients With Glenohumeral Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sibel Gayretli Atan, Physiotherapist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ''IU''
Record Dates: First submitted 2019-04-11; First posted 2019-05-21 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-11

CONDITIONS: Glenohumeral Arthritis
Keywords: Glenohumeral Arthritis; Pain; Mobilisation; Physiotherapy; Rehabilitation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ''Manuel Therapy group'' (Experimental): This treatment group will be received Manuel Therapy techniques and exercise interventions.
  Interventions: Other: Manuel Therapy plus Exercise Intervention
- ''Exercise group'' (Experimental): This treatment group will be received only exercise interventions.
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Manuel Therapy plus Exercise Intervention — Shoulder mobilization techniques include glenohumeral traction, anterior, posterior and inferior glide. We will also use anterior, posterior and inferior joint stretching exercises and scapular mobilization. Exercise interventions include range of motion exercises, stretching exercises, strengthening exercises, and pendulum exercises.
  Arms: ''Manuel Therapy group''
Other: Exercise Intervention — Exercise interventions include range of motion exercises, stretching exercises, strengthening exercises, and pendulum exercises.
  Arms: ''Exercise group''

SUMMARY:
The aim of the investigator's study is to compare the efficacy of manual therapy and exercise practices compared to exercise practice in patients with Glenohumeral Arthritis. Thirty volunteer patients will include into the study.

DETAILED DESCRIPTION:
Patients will randomly divide into two groups. A common exercise program was applied to both groups during 15 sessions. Manual therapy techniques will apply to the manual therapy group in addition to exercise practices. Patients will evaluate in terms of functional status, pain, range of motion, muscle strength and health-related quality before and after 5 weeks of treatment. Also, patient's satisfaction from treatment will evaluate at the 5th week of the treatment. DASH and ASES forms for functional status, VAS for pain, digital goniometer for range of motion, manual muscle test for muscle strength, SF-12 for health-related quality of life, and Global Rating of Change (GRC) Scale for patient satisfaction will be used as evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older patients
* To be diagnosed with GHOA by specialist physician via MRI, US or radiography and physical examination
* Unilateral shoulder pain lasting more than 2 months seen during daily living activities and at rest

Exclusion Criteria:

Patients with:

* Severe arthrosis
* Tumor
* Cervical radiculopathy
* Emotional or cognitive problems
* A neurological disease that causes muscle weakness on the shoulder
* A skin disease that may affect upper extremity assessment.
* Frozen shoulder
* Thoracic outlet syndrome

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of Motion (ROM) | Evaluation will be performed first time at baseline and second time will be performed after 5 weeks rehabilitation program. After treatment "change" will be assessed.
  The shoulder flexion, abduction, internal and external rotation ROM will be evaluated with digital goniometer while the patient will be in supine position.

SECONDARY OUTCOMES:
ASES (The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment) Form | Evaluation will be performed before treatment and after 5 weeks rehabilitation program.
  ASES is an assessment form prepared by shoulder and elbow surgeons with objective and subjective sections. The total score is at least 0 and at most 100, and the high scores are positively correlated with the normal function.
Visual Analogue Scale (VAS) | Evaluation will be performed before treatment and after 5 weeks rehabilitation program.
  The levels of pain is felted at rest / activity / night will be measured using Visual Analogue Scale (VAS).Patients will be asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain.
Manual Muscle Test | Evaluation will be performed before treatment and after 5 weeks rehabilitation program.
  Manual Muscle Test is a procedure for the evaluation of strength of individual muscle or muscles group, based upon the effective performance of a movement in relation to the forces of gravity or manual resistance through the available ROM.
Short Form 12 (SF-12) | Evaluation will be performed before treatment and after 5 weeks rehabilitation program.
  SF-12 will be used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with high quality of life.
Global Rating of Change (GRC) Scale | Evaluation will be performed after 5 weeks rehabilitation program.
  Global Rating of Change (GRC) scale will be used to assess the overall satisfaction levels of the patients. Patients will be asked to evaluate their post-treatment status with a 5-point likert scale and high scores are positively correlated with satisfaction.
The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Evaluation will be performed before treatment and after 5 weeks rehabilitation program.
  DASH questionnaire inquires about the activities of a person in daily life, the degree of participation in recreational activities, the symptom and psychosocial state that affects their pain, emotional state and sleep quality. The total score is at least 0 and at most 100, and the high scores are positively correlated with the increased functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Gayretli Atan, Principal Investigator — sssibel_38@hotmail.com
Locations (1):
- Istanbul University, Bakırköy, Istanbul, Turkey (Türkiye)